CLINICAL TRIAL: NCT03898349
Title: Evaluation of the Initial Deployment of VA's Annie Texting System (PEC 15-470)
Brief Title: eHealth Partnered Evaluation Initiative - Evaluation of the Initial Deployment of VA's Annie Texting System
Acronym: AnnieEval
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Office of Connected Care (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: PEX 19-001
Record Dates: First submitted 2019-03-20; First posted 2019-04-02 (Actual); Results first posted 2019-12-13 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Hepatitis C
Keywords: Automated Text Messaging System; Implementation science; Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Intervention Model Description: Four facilities were randomized to serve as intervention sites and receive our augmented implementation strategy. These facilities had regular facilitation calls, a site visit to assist with implementation, and were given the toolkit, in addition to receiving usual implementation assistance. An additional three comparison sites received usual implementation of Annie only, which involves an orientation/training meeting and the option of attending twice-monthly Annie clinical adoption calls run by the Office of Connected Care. Two control sites did not receive Annie.
Who Masked: Participant, Care Provider
Masking Description: Patients and providers did not know which facilitation group they were in
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-Texters (No Intervention): Patients did not receive the automated text messaging system "Annie"
- Texters (Active Comparator): Patients received the Annie text messaging system for patient self-management of HCV treatment including medication, lab, and appointment reminders, and motivational messages.
  Interventions: Other: Annie text messaging system; Other: Annie text messaging system with Usual implementation; Other: Annie text messaging system with Augmented implementation

INTERVENTIONS:
Other: Annie text messaging system — Annie text messaging system for patient self-management of HCV treatment including medication, lab, and appointment reminders, and motivational messages.
  Arms: Texters
Other: Annie text messaging system with Usual implementation — Three comparison sites received usual implementation of the automated text messaging system "Annie" only, which involves an orientation/training meeting and the option of attending twice-monthly Annie clinical adoption calls
  Arms: Texters
Other: Annie text messaging system with Augmented implementation — Four facilities received the automated text messaging system "Annie" and our augmented implementation strategy. These facilities had regular facilitation calls, a site visit to assist with implementation, and were given the toolkit, in addition to receiving usual implementation assistance
  Arms: Texters

SUMMARY:
Conduct a rigorous formative evaluation of the initial deployment of the Annie texting system across several pilot test sites and from these findings, develop and test an augmented implementation strategy to facilitate more rapid adoption of Annie across VA.

DETAILED DESCRIPTION:
The investigators examined patient and provider experiences with VA's automated text messaging system, named "Annie". The investigators aimed to describe early experiences using Annie and subsequently pilot and evaluate an augmented implementation strategy to improve implementation of the system. Then, seven new facilities implemented Annie. The investigators focused on specialty clinics serving patients with hepatitis-C virus (HCV). Working in collaboration with clinical team members and other Office of Connected Care stakeholders, the investigators developed a texting protocol for Veterans with HCV that included motivational messages, medication and lab appointment reminders. This protocol was made available to the seven new facilities. Four facilities were randomized to serve as intervention sites to receive augmented implementation strategy. These facilities had regular facilitation calls, a site visit to assist with implementation, and were given the toolkit, in addition to receiving usual implementation assistance, described below. An additional three comparison sites received usual implementation of Annie only, which involves an orientation/training meeting and the option of attending twice-monthly Annie clinical adoption calls run by the Office of Connected Care. Two control sites did not receive Annie. The investigators conducted a mixed-methods evaluation including pre and post patient and provider surveys and semi-structured interviews, medical chart abstraction, and process measure analysis. The investigators collected data on patient and clinician experiences with the Annie system, including usability, clinical workflow fit, and clinical benefits such as improved HCV medication adherence and rates of appropriately timed lab tests.

ELIGIBILITY:
Inclusion Criteria:

* Starting HCV treatment at a VA clinic
* Have access/ability to text messaging

Exclusion Criteria:

* Not being treating for HCV
* No access/ability to use a cell phone

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Patrick Hogan, PhD MS BS, Principal Investigator — VA Bedford HealthCare System, Bedford, MA; Christopher Gillespie, PhD MA BS, Principal Investigator — VA Bedford HealthCare System, Bedford, MA; Donald K McInnes, ScD MS BA, Principal Investigator — VA Bedford HealthCare System, Bedford, MA
Locations (1):
- VA Bedford HealthCare System, Bedford, MA, Bedford, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yakovchenko V, McInnes DK, Petrakis BA, Gillespie C, Lipschitz JM, McCullough MB, Richardson L, Vetter B, Hogan TP. Implementing Automated Text Messaging for Patient Self-management in the Veterans Health Administration: Qualitative Study Applying the Nonadoption, Abandonment, Scale-up, Spread, and Sustainability Framework. JMIR Mhealth Uhealth. 2021 Nov 15;9(11):e31037. doi: 10.2196/31037. PMID 34779779
- [Derived] Yakovchenko V, Hogan TP, Houston TK, Richardson L, Lipschitz J, Petrakis BA, Gillespie C, McInnes DK. Automated Text Messaging With Patients in Department of Veterans Affairs Specialty Clinics: Cluster Randomized Trial. J Med Internet Res. 2019 Aug 4;21(8):e14750. doi: 10.2196/14750. PMID 31444872

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was not an intent to treat design, therefore UI and AI groups were combined to compare texters and non-texters from each of the groups (and control).
Groups:
- Non-texters: Patients who did not receive the automated text messaging system "Annie"
- Texters: Patients who did receive the automated text messaging system "Annie"
  Annie text messaging system: Annie text messaging system for patient self-management of HCV treatment including medication, lab, and appointment reminders, and motivational messages.
  Annie text messaging system with Usual implementation: Three comparison sites received usual implementation of the automated text messaging system "Annie" only, which involves an orientation/training meeting and the option of attending twice-monthly Annie clinical adoption calls
Period: Overall Study
Arm/Group | Non-texters | Texters
Started | 125 | 625
Completed | 15 | 15
Not Completed | 110 | 610

BASELINE CHARACTERISTICS:
Population: "Non-texters" could come from UI or AI clinics (patients who agreed to participate in the project but never completed the last step of authenticating themselves with the aTS, and thus never received any text messages), as well as from the two comparison clinics that did not implement the aTS. "Texter" could come from either UI or AI clinics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-Texters | Texters | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The 30 are those in the 2 arms who were analyzed.
  years | 62 (11) | 62 (6) | 62 (11)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: we did not have demographic characteristics for the overall population
  Participants
    Female | 1 | 1 | 2
    Male | 14 | 14 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — The 30 are those in the 2 arms who were analyzed.
  Participants
    African American or Black | 6 | 13 | 19
    White | 8 | 2 | 10
    Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Perception of HCV Treatment Success
Description: The primary goal of the automated text messaging system is to improve patient self-management. As such, we measured illness perception and patient activation using a validated instrument adapted for HCV (Fisher L, Glasgow RE, Mullan JT, Skaff MM, Polonsky WH. Development of a brief diabetes distress screening instrument. Ann Fam Med 2008;6(3):246-252). The item "Feeling that I am failing with my HCV treatment" represents patient perceptions about their ability to take medications as prescribed and reflects concerns about failing HCV treatment.
Time Frame: Post (after 12 weeks of Annie text messaging use)
Population: This was not an intent to treat design, therefore UI and AI groups were combined to compare texters and non-texters from each of the groups (and control).
Measure: Count of Participants; unit: Participants
Groups:
- Non-texters: Patients who did not receive Annie text messages
  Annie text messaging system: Annie text messaging system for patient self-management of HCV treatment including medication, lab, and appointment reminders, and motivational messages.
  Annie text messaging system with Usual implementation: Three comparison sites received usual implementation of the automated text messaging system "Annie" only, which involves an orientation/training meeting and the option of attending twice-monthly Annie clinical adoption calls
- Texters: Patients who received Annie text messages
  Annie text messaging system: Annie text messaging system for patient self-management of HCV treatment including medication, lab, and appointment reminders, and motivational messages.
  Annie text messaging system with Augmented implementation: Four facilities received the automated text messaging system "Annie" and our augmented implementation strategy. These facilities had regular facilitation calls, a site visit to assist with implementation, and were given the toolkit, in addition to receiving usual implementation assistance
Arm/Group | Non-texters | Texters
Number analyzed (Participants) | 15 | 15
Participants | 8 | 13

ADVERSE EVENTS:
Time Frame: 1 year
Description: Definition is consistent with clinicaltrials.gov
Groups:
- Non-texters: Patients who did not receive Annie text messages for patient self-management of HCV treatment including medication, lab, and appointment reminders, and motivational messages.
- Texters: Patients who did receive Annie text messages for patient self-management of HCV treatment including medication, lab, and appointment reminders, and motivational messages.
Arm/Group | Non-texters | Texters
All-Cause Mortality (participants affected / at risk) | 0/125 | 0/625
Serious Adverse Events (participants affected / at risk) | 0/125 | 0/625
Other Adverse Events (participants affected / at risk) | 0/125 | 0/625

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-10): https://cdn.clinicaltrials.gov/large-docs/49/NCT03898349/Prot_SAP_000.pdf